CLINICAL TRIAL: NCT04252079
Title: Endovascular Repair of Juxtarenal Aortic Aneurysm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Mohamed Awad Hassan, Assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Aortic aneurysm repair
Record Dates: First submitted 2020-01-18; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Juxtarenal Aortic Aneurysm

STUDY DESIGN:
Intervention Model Description: Prospective cross sectional study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- We compare different endovascular techniques as an alternative (Other): We compare different endovascular techniques as an alternative to surgical reconstruction to repair JAAS regarding ; success rates, 30-day mortality, endoleak events secondary intervention rates
  Interventions: Procedure: Endovascular Repair of Juxtarenal Aortic Aneurysm

INTERVENTIONS:
Procedure: Endovascular Repair of Juxtarenal Aortic Aneurysm — 1. History taking and clinical examination.
  2. Preoperative Imaging
     CTA is the cross-sectional imaging modality of choice.
  3. Preoperative evaluation
     a-Renal evaluation
     b_ cardiac evaluation C-Pulmonary evaluation
  4. Surgical techniques
     1. Anesthesia The use of general anesthesia due to the duration of the procedures and the necessity to control patient breathing to allow precise imaging and accurate device deployment.
     2. Intra operative imaging A "hybrid" operating room with high-quality fixed imaging is needed for the performance of FEVAR.
  C-Device delivery and deployment all FEVAR procedures begin with access of the femoral arteries by either open or percutaneous technique.

SUMMARY:
The investigators compare different endovascular techniques as an alternative to surgical reconstruction to repair JAAS regarding ; success rates, 30-day mortality,endoleak events secondary intervention rates

DETAILED DESCRIPTION:
Aortic disease is the direct cause of close to 10000 deaths annually in the United States. 1

Aneurysmal disease can affect any segment of the aorta, from the aortic root to the aortic bifurcation. Juxtarenal Aortic Aneurysms (JAA) (where a specialty designed custom -made device (endograft)which has holes, or fenestrations ,on the graft body to maintain the patency of the visceral arteries) account for approximately 15% of abdominal aortic aneurysms.2

Successful aortic aneurysm treatment depends on either open replacement or endovascular exclusion of the aneurysmal segment with healthy artery proximal and distal to the repair.

The decision to treat an AAA is based on the associated risk of treatment, the risk of aneurysm rupture, the patient's life expectancy, and patient preference.

The primary determinant of rupture risk is maximum aneurysm diameter, with negligible rupture risk in aneurysms <4cm in diameter compared with aneurysms >8 cm . 3, 4.

The Society for Vascular Surgery recommends repair for all patients of acceptable perioperative risk with an AAA ≥5.5 cm in diameter as well as all patients with saccular and symptomatic aneurysms.5 ,6

These guidelines also suggest repair for women at a diameter of 5.0 cm.

Fenestrated Endovascular Aneurysm Repair (FEVAR) and Chimney Endovascular Aneurysm Repair (CHEVAR)are both effective methods to treat JAAs

ELIGIBILITY:
Inclusion Criteria:

* • Subject is ≥18 years old

  * Subject is scheduled for treatment of the juxtarenal aortic aneurysm with a short infrarenal neck aortic neck length <15 mm, neck angulation >60%, conical neck) (i.e. denovo cases).
  * Subject is able and willing to comply with the protocol and to adhere to the follow-up requirements.
  * Subject has provided written informed consent.

Exclusion Criteria:

* Subject is participating in a concurrent study which may confound study results

  * Subject has a life expectancy ≤1 year
  * Subject has an aneurysm that is:

    * Mycotic
    * Inflammatory
    * Pseudoaneurysm
  * Subject requires emergent aneurysm treatment, for example, trauma or rupture
  * Subject has previously undergone surgical treatment for abdominal aortic aneurysm
  * Subject is a female of childbearing potential in whom pregnancy cannot be excluded
  * Subject has a known hypersensitivity or contraindication to anticoagulants, anti-platelets, or contrast media, which is not amenable to pre-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be clinical success . | One year
  Clinical success will be evaluated by Measurment of blood pressure by sphygmomanometer in mmhg Serum creatinine level in mg/dL
One year patency of the endovascular graft | One year
  One year patency will be assessed by CT angiography ( if it is patent or not).
  CT angiography can detect successful deployment of the endovascular device at the intended location or post endograft complications as type I or III endoleak , graft thrombosis, aneurysm expansion , aneurysm rupture.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf G Taha, MD, Study Director — Assistant professur Assiut University

REFERENCES:
- [Background] Taylor SM, Mills JL, Fujitani RM. The juxtarenal abdominal aortic aneurysm. A more common problem than previously realized? Arch Surg. 1994 Jul;129(7):734-7. doi: 10.1001/archsurg.1994.01420310066011. PMID 8024454
- [Background] Brown LC, Powell JT. Risk factors for aneurysm rupture in patients kept under ultrasound surveillance. UK Small Aneurysm Trial Participants. Ann Surg. 1999 Sep;230(3):289-96; discussion 296-7. doi: 10.1097/00000658-199909000-00002. PMID 10493476
- [Background] Chaikof EL, Dalman RL, Eskandari MK, Jackson BM, Lee WA, Mansour MA, Mastracci TM, Mell M, Murad MH, Nguyen LL, Oderich GS, Patel MS, Schermerhorn ML, Starnes BW. The Society for Vascular Surgery practice guidelines on the care of patients with an abdominal aortic aneurysm. J Vasc Surg. 2018 Jan;67(1):2-77.e2. doi: 10.1016/j.jvs.2017.10.044. PMID 29268916
- [Background] Moll FL, Powell JT, Fraedrich G, Verzini F, Haulon S, Waltham M, van Herwaarden JA, Holt PJ, van Keulen JW, Rantner B, Schlosser FJ, Setacci F, Ricco JB; European Society for Vascular Surgery. Management of abdominal aortic aneurysms clinical practice guidelines of the European society for vascular surgery. Eur J Vasc Endovasc Surg. 2011 Jan;41 Suppl 1:S1-S58. doi: 10.1016/j.ejvs.2010.09.011. No abstract available. PMID 21215940
- [Background] Greenberg R, Eagleton M, Mastracci T. Branched endografts for thoracoabdominal aneurysms. J Thorac Cardiovasc Surg. 2010 Dec;140(6 Suppl):S171-8. doi: 10.1016/j.jtcvs.2010.07.061. PMID 21092788
- [Background] Coselli JS, LeMaire SA, Preventza O, de la Cruz KI, Cooley DA, Price MD, Stolz AP, Green SY, Arredondo CN, Rosengart TK. Outcomes of 3309 thoracoabdominal aortic aneurysm repairs. J Thorac Cardiovasc Surg. 2016 May;151(5):1323-37. doi: 10.1016/j.jtcvs.2015.12.050. Epub 2016 Jan 14. PMID 26898979
- [Background] Eagleton MJ, Follansbee M, Wolski K, Mastracci T, Kuramochi Y. Fenestrated and branched endovascular aneurysm repair outcomes for type II and III thoracoabdominal aortic aneurysms. J Vasc Surg. 2016 Apr;63(4):930-42. doi: 10.1016/j.jvs.2015.10.095. Epub 2016 Jan 11. PMID 26792544